CLINICAL TRIAL: NCT04953195
Title: Effect of Thyroid Replacement Therapy on Thyroid Structure in Patients With Subclinical Hypothyroidism
Brief Title: Thyroid Replacement Therapy in Patients With Subclinical Hypothyroidism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Director of Endocrinology, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-309
Record Dates: First submitted 2021-06-25; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Subclinical Hypothyroidisms
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- levothyroxine sodium (Experimental): levothyroxine sodium
  Interventions: Drug: Levothyroxine Sodium Tablets

INTERVENTIONS:
Drug: Levothyroxine Sodium Tablets — Levothyroxine Sodium(50ug/Tablets,dosage form 25ug,once a day) was administered to patients with autoimmune thyroiditis with mild subclinical hypothyroidism,

SUMMARY:
The purpose of this experiment is to compared the changes of thyroid function, anti-thyroid peroxidase antibody, anti-thyroglobulin antibody, thyroid magnetic resonance T1-mapping and various metabolic indexes from baseline to the end of treatment (after the thyroid function had been normal for more than three months)

DETAILED DESCRIPTION:
In patients with autoimmune thyroiditis with mild subclinical hypothyroidism, the study period will include a screening period of not more than 30 days, and a 12-week treatment period compared to baseline. At completion of treatment, Thyroid Stimulating Hormone(TSH), free thyroxine (FT4)，free thyroxine (FT3) will be included. The changes of anti-thyroglobulin antibody, anti-thyroglobulin antibody, T1-mapping and metabolic indexes.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 18 and 75;
* Diagnostic criteria for mild subclinical hypothyroidism :TSH>10mIU/L, thyroxine and free thyroxine levels were normal
* Positive thyroglobulin antibody and/or Thyroperoxidase antibody
* No previous use of drugs affecting thyroid function

Exclusion Criteria:

* The contraindications indicated in the Chinese instructions of the drug
* Liver function impairment
* Renal function impairment
* Claustrophobia
* Mental disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Thyroid Stimulating Hormone changes | Thyroid Stimulating Hormone Changes from baseline and 12 weeks during follow-up
  Thyroid Stimulating Hormone Changes from baseline and 12 weeks during follow-up
free thyroxine changes | free thyroxine changes from baseline and 12 weeks during follow-up
  free thyroxine changes from baseline and 12 weeks during follow-up
T1-mapping values of Thyroid MRI | T1-mapping values of Thyroid MRI Changes from baseline and 12 weeks during follow-up
  T1-mapping values of Thyroid MRI Changes from baseline and 12 weeks during follow-up
Free triiodothyronine changes | Free triiodothyronine changes Changes from baseline and 12 weeks during follow-up
  Free triiodothyronine changes Changes from baseline and 12 weeks during follow-up

SECONDARY OUTCOMES:
anti-thyroid peroxidase antibody changes | anti-thyroid peroxidase antibody changes from baseline and 12 weeks during follow-up
  anti-thyroid peroxidase antibody changes from baseline and 12 weeks during follow-up
anti-thyroglobulin antibody changes | anti-thyroglobulin antibody changes from baseline and 12 weeks during follow-up
  anti-thyroglobulin antibody changes from baseline and 12 weeks during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, MD, Principal Investigator — Beijing Chao-Yang Hospital, Capital Medical University, Beijing
Locations (1):
- Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China